CLINICAL TRIAL: NCT04449224
Title: Comparative Effectiveness of Biologic Disease-modifying Antirheumatic Drugs and Small Molecular Inhibitors in Patients With Moderate to Severe RA: Prospective Observational Study
Brief Title: Comparative Effectiveness of Targeted Therapy in RA Patients
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Hanyang University (Other)
Collaborators: Ministry of Health, Republic of Korea (Other Government)
Responsible Party: Principal Investigator, Yoon-Kyoung Sung, Principal Investigator, Hanyang University
Other Study IDs: HUHRD-SPE-20-01
Record Dates: First submitted 2020-06-07; First posted 2020-06-26 (Actual); Last update posted 2020-06-26 (Actual); Status verified 2020-06

CONDITIONS: Rheumatoid Arthritis
Keywords: Arthritis; Arthritis, Rheumatoid; Joint Diseases; Musculoskeletal Diseases
MeSH Terms: conditions — Arthritis, Rheumatoid; Arthritis; Joint Diseases; Musculoskeletal Diseases | interventions — Etanercept; tocilizumab; Abatacept; Adalimumab; tofacitinib; baricitinib

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 48 Weeks
Biospecimen Retention: Samples Without DNA — Serum (restricted to a patient who provides written consent to biosampling)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- RA patients who start bDMARD: The efficacy and safety of targeted therapy will be evaluated in RA patients who are treated with a biologic disease modifying antirheumatic drug (bDMARD) including Adalimuab, Etanercept, Tocilizumab or Abatacept after shared-decision making.
  Interventions: Drug: Adalimuab, Etanercept, Tocilizumab, or Abatacept
- RA patients who start small molecule inhibitor: The efficacy and safety of targeted therapy will be evaluated in RA patients who are treated with a small molecular inhibitor including Tofacitinib or Baricitinib after shared-decision making.
  Interventions: Drug: Tofacitinib or Baricitinib

INTERVENTIONS:
Drug: Adalimuab, Etanercept, Tocilizumab, or Abatacept — A specific targeted therapy wil be decided by shared-decision making, a bidirectional process in which clinicians and patients make decisions based on clinical evidence that balances risks and expected outcomes with patient preferences and values.
  Other Names: Humira, Enbrel, Etoloche, Eucept, Actemra, or Orencia
  Groups: RA patients who start bDMARD
Drug: Tofacitinib or Baricitinib — A specific targeted therapy wil be decided by shared-decision making, a bidirectional process in which clinicians and patients make decisions based on clinical evidence that balances risks and expected outcomes with patient preferences and values.
  Other Names: Xeljanz or Olumiant
  Groups: RA patients who start small molecule inhibitor

SUMMARY:
The objective of a multicenter prospective observational study is to compare effectiveness and safety of biologic disease-modifying antirheumatic drugs and small molecular inhibitors in patients with moderately to severely active rheumatoid arthritis patients who have had an inadequate response or intolerace to methotrexate.

DETAILED DESCRIPTION:
This study is a multicenter prospective observational study to show non-inferiority of clinical efficacy for small molecular inhibitors after 48 week of treatment to biologic disease modifying anti-rheumatic drugs (bDMARDs) in patients having moderately to severely active RA and who have been intolerant to conventional synthetic disease modifying anti-rheumatic drugs (csDMARDs) including methotrexate.

Primary end point is a percentage of participants of achieving low disease activity according to Disease Activity Score in 28 joints-Erythrocyte Sedientation Rate (DAS28-ESR) at weeks 24. A total of 506 RA patients will be included, and allocated in ratio of 1:1 to bDMARD group and small molecule inhibitor group. Group allocation is determined by shared-decision making, so that the number of participants could be re-assessed according to recruitment status of participatns.

ELIGIBILITY:
Inclusion Criteria:

Patients are included in this study if they are:

* 19 years or olders
* Patients who satisfy the 1987 American College of Rheumatology (ACR) or 2010 American College of Rheumatology/European League Against Rheumatism (ACR/EULAR) classification criteria for RA
* Patients having moderately to severely active RA who are intolerant to csDMARDs including methotrexate and those who have never been exposed to bDMARDs or small molecular inhibitors before
* Patients who provide written consent to participate in this study

Exclusion Criteria:

* Patients who are contraindicated to bDMARDs or small molecule inhibitor
* Patients who have plans for pregnancy or elective surgery
* Patients who had ever diagnosed with any malignancy or are treated for malginancy
* Patients who cannot voluntarily provie a written consent to participate in this study
* Patients who did not provide a written consent to participate in this study

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Korean RA patients who start biologic disease modifying anti-rheumatic drugs (bDMARDs) or small molecule inhibitors with moderately to severely active RA who have had an inadequate response or intolerance to methotrexate and naive to any bDMARDs or small molecule inhibitors.
Sampling Method: Non-Probability Sample
Enrollment: 506 (Estimated)
Dates: Start 2020-04-27 (Actual); Primary Completion 2023-08-19 (Estimated); Study Completion 2024-08-19 (Estimated)

PRIMARY OUTCOMES:
Percentage of participants achieving low disease activity according to Disease Activity Score 28 joints-Erythrocyte sedimentation (DAS28-ESR) | At weeks 24
  Disease Activity Score 28 joints-Erythrocyte sedimentation (DAS28-ESR) below 3.2 indicates low disease activity of RA.

SECONDARY OUTCOMES:
Changes in Health Assessment Questionnaire (HAQ) | At weeks 12, 24, and 48
  The HAQ-DI is a patient-reported assessment of physical function that includes 20 items in eight categories representing a comprehensive set of functional activities, including dressing and grooming, arising, eating, walking, hygiene, reach, grip and common daily activities. Patients are asked about their ability to complete these tasks in the past week using the following categories: without any difficulty (0); with some difficulty (1); with much difficulty (2); and unable to do (3). Scores on each task were summed and averaged to provide an overall score ranging from 0 (best) to 3 (worst), with a higher score representing a high-dependency disability.
Changes in EuroQol-5 dimension (EQ-5D) | At weeks 12, 24, and 48
  The EQ-5D is a generic instrument for measuring health-related quality of life. The EQ-5D-5L essentially consists of two parts: the EQ-5D descriptive system and the EQ visual analogue scale (EQ VAS). Patients are asked about their ability to complete specific tasks today using the following dimensions: mobility, self-care, usual activities, pain/discomfort and anxiety/depression. Each dimension has 5 levels: no problems (1), slight problems (2), moderate problems (3), severe problems (4) and extreme problems (5). EQ-5D-5L health states can be summarised using the 5-digit code, after that, it is represented by a single summary number (index scores). Health state index scores generally range from less than 0 (where 0 is the value of a health state equivalent to dead; negative values representing values as worse than dead) to 1 (the value of full health), with higher scores indicating higher health utility.
Changes in EuroQol visual analogue scale (EQ VAS) | At weeks 12, 24, and 48
  The EQ-5D is a generic instrument for measuring health-related quality of life. The EQ-5D-5L essentially consists of two parts: the EQ-5D descriptive system and the EQ visual analogue scale (EQ VAS). The second part of the questionnaire consists of a visual analogue scale (VAS) on which the patient rates his/her perceived health from 0 (the worst imaginable health) to 100 (the best imaginable health).
Percentage of participants achieving low disease activity according to Disease Activity Score 28 joints-Erythrocyte sedimentation rate (DAS28-ESR) | At weeks 12 and 48
  Disease Activity Score 28 joints-Erythrocyte sedimentation (DAS28-ESR) below 3.2 indicates low disease activity of RA.
Percentage of participants achieving remission according to Disease Activity Score 28 joints-Erythrocyte sedimentation rate (DAS28-ESR) | At weeks 12, 24, and 48
  Disease Activity Score 28 joints-Erythrocyte sedimentation (DAS28-ESR) below 2.6 indicates remission of RA.
Percentage of participants with European League Against Rheumatism (EULAR) Response according to Disease Activity Score 28 joints-Erythrocyte sedimentation rate (DAS28-ESR) | At weeks 12, 24, and 48
  The European League Against Rheumatism (EULAR) response criteria classify patients as good, moderate, or nonresponders, using the individual amount of change in DAS28 and the level of DAS reached (low, moderate, or high); good responders were patients with an improvement of >1.2 and a present score of ≤3.2; moderate responders were patients with an improvement of >0.6 to ≤1.2 and a present score of ≤5.1, or an improvement of >1.2 and a present score of >3.2; non-responders were any patients with an improvement of ≤0.6, or patients with an improvement of >0.6 to 1.2 and a present score of >5.1
Percentage of participants having radiologic progression in RA (if possible) | At weeks 48
  Percentage of participants having radiologic progression in rheumatoid arthritis (if possible)
Percentage of participants having changes in ultrasonographic findings of RA (if possible) | At weeks 48
  Percentage of participants having changes in ultrasonographic findings of rheumatoid arthritis (if possible)
Biomarkers predictive of treatment response of RA (if possible) | At weeks 24
  We would like to discover serum biomarkers predicting 24-week treatment response in each targeted therapy for RA patients. Serum samples will be collected before target therapies (at 0 week) and grouped according to the treatment response after 24 weeks. The putative biomarkers predicting treatment response will be screened using proteomics method and validated via ELISA.
Incidence of adverse events (AEs) or serious adverse events (SAEs) of targeted therapy (if possible) | At weeks 48
  Incidence of adverse events (AEs) or serious adverse events (SAEs) of targeted therapy (if possible)
Compliance with targeted therapy defined by Patient-reported adherence and Modified Morisky scale (if possible) | At weeks 48
  This 6-item questionnaire measures two domains of adherence; knowledge and motivation. Patients are categorized as having 'high' or 'low' knowledge and motivation based on their yes or no response to each of the six questions of the Modified Morisky Scale. Each 'no' response to each question results in +1 (except question 5, in which a 'yes' response would result in +1) and 'yes' responses to each question result in +0 (except question 5, where a 'no' response would result in +0). Scores for the 6-item of Modified Morisky Scale can range from 0 to 6, with higher scores indicating better adherence.

CONTACTS AND LOCATIONS:
Overall Officials: Yoon-Kyoung Sung, MD, PhD, MPH, Principal Investigator — Hanyang University
Locations (1):
- Hanyang University, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No